CLINICAL TRIAL: NCT04016506
Title: Retrospective and Prospective Study on the Epidemiology, Management and Complications Related to Pancreatic Trauma in Children
Brief Title: Epidemiology, Management and Complications Related to Pancreatic Trauma in Children
Acronym: PANC-TRAUMA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/18OCT/394
Record Dates: First submitted 2019-07-09; First posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Pancreas Injury; Child, Only
Keywords: Pancreas Injury; Child

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pancreas injury: children with Pancreas trauma
  Interventions: Other: nutritional questionnaire

INTERVENTIONS:
Other: nutritional questionnaire — nutritional questionnaire is given to the patient after the injury

SUMMARY:
The aim of this study is to better evaluate the treatment and development of children and adolescents who have had a pancreatic trauma and who are being followed in Belgian hospitals.

DETAILED DESCRIPTION:
The aim of this study is to better evaluate the treatment and development of children and adolescents who have had a pancreatic trauma and who are being followed in Belgian hospitals.

Through this study, the investigators hope to be able to understand:

1. The epidemiology of pancreatic trauma in Belgium. How these traumas occur (accident, fall,...).
2. Pancreatic trauma management in Belgian hospitals according to severity grade.
3. Short- and medium-term complications associated with the trauma
4. Long-term complications of trauma on growth and on the endocrine and exocrine function of the pancreas.

On the basis of all the information collected, the investigators hope to be able to provide indicators on the epidemiology of pancreatic trauma in children, short-term risks as well as nutritional and functional risks, taking into account the initial management of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Child aged ˂18 years at the time of the trauma
* Child regularly followed in paediatric gastroenterology consultation
* Positive history of pancreatic trauma
* Child with at least one blood lipase measurement
* Child with at least one pancreatic imaging available

Exclusion Criteria:

* age >18 years

Max Age: 17 Years | Sex: All
Age Groups: Child
Study Population: * Child aged ˂18 years at the time of the trauma
  * Child regularly followed in paediatric gastroenterology consultation
  * Positive history of pancreatic trauma
  * Child with at least one blood lipase measurement
  * Child with at least one pancreatic imaging available
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-09-15 (Estimated); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
incidence of pancreas injury in children | from start of inclusion to 2 years thereafter
  number of new diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Scheers, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (3):
- Belgium (3):
  - Cliniques universitaires Saint-Luc, Brussels
  - Erasme/HUDERF, Brussels
  - ULG La Citadelle, Liège

IPD SHARING:
Plan to Share IPD: No